CLINICAL TRIAL: NCT07044245
Title: Evaluation of the Effect of Low Level Diode Laser Biostimulation on Implant Stability in Immediate Implant in The Maxillary Premolars. A Randomized Clinical Trial.
Brief Title: Effect of Low Level Diode Laser Biostimulation on Implant Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLLT-premolars
Record Dates: First submitted 2025-06-19; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Immediate Implant Placement; Laser; Biostimulation
Keywords: immediate implant; ISQ; LLLT; clinical stability

STUDY DESIGN:
Intervention Model Description: Patients with immediate implant placement in the of maxillary premolars with low laser Biostimulation
Who Masked: Participant, Outcomes Assessor
Masking Description: Sequentially numbered, opaque, sealed envelopes (SNOSE) allocation concealment method will be utilized. Each participant included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each participant is allocated and placed inside opaque envelopes carrying the respective names of participants. A trial independent personnel will be assigned the role of keeping the envelopes and unfolding them only at the time of the operation, so that the participant is allocated to a group which is concealed from the operator Furthermore, outcome assessor was blinded from the group enrollment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with immediate implant placement in maxillary premolars receiving low laser Biostimulation (Active Comparator): Patients with immediate implant placement in maxillary premolars receiving low laser Biostimulation after placement on two sessions
  Interventions: Procedure: immediate maxillary premolar implant placement with subsequent laser Biostimulation
- Patients with immediate implant placement in maxillary premolars receiving sham laser (Sham Comparator): Patients with immediate implant placement in maxillary premolars receiving sham laser as a control
  Interventions: Procedure: immediate maxillary premolar implant placement with no subsequent laser Biostimulation

INTERVENTIONS:
Procedure: immediate maxillary premolar implant placement with no subsequent laser Biostimulation — Sham laser application
  Arms: Patients with immediate implant placement in maxillary premolars receiving sham laser
Procedure: immediate maxillary premolar implant placement with subsequent laser Biostimulation — low lever biostimulation was performed on two consecutive sessions each of 100 s. First session was carried out immediately on surgery time after implant placement, using a diode laser Photo-biomodulation tip in a continuous wave and non-contact mode
  Arms: Patients with immediate implant placement in maxillary premolars receiving low laser Biostimulation

SUMMARY:
Tooth loss is accompanied by bone loss in all dimensions, so preservation of the bone is mandatory for placement of dental implant, as bone quantity and quality are predictive factors in achieving proper primary stability. Low level bio stimulation has stimulatory effect on bone cells so it can be used in immediate implants to increase bone formation around the implant.

the Aim of this study is to evaluate the effect of low-level diode laser Biostimulation on immediate implants in maxillary premolars.

DETAILED DESCRIPTION:
20 patients with unrestorable maxillary premolars were included in the study treated with immediate implants. Patients were divided into two groups (n=10). Group 1 Received immediate implant with low level diode laser application (study), and group 2 received immediate implant without laser application (control). Preoperative clinical and radiographic evaluation, immediate post operative and after 4 months radiographic evaluation to assess stability and bone density around the implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unrestorable maxillary premolars with sufficient bone quantity to receive the dental implant.
2. Age ranging from 25-45.
3. Patients with no local or systemic pathology that can interfere with normal wound healing.
4. Non- smokers.
5. Patients that are properly motivated to complete follow up visits.
6. Patients with adequate oral hygiene or willing to improve their oral hygiene to ensure uncompromised wound healing.

Exclusion Criteria:

1. Patients with uncontrolled medical condition that can affect surgical outcome or bone and wound healing. (ex: diabetes mellitus)
2. Patients with periapical pathology that may contraindicate immediate implant placement.
3. History of receiving irradiation in head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Implant Stability Assessment using Radio frequency analysis | 4 month
  Secondary implant stability analysis was performed 4-months after implant placement. Radio frequency analysis (RFA) was performed using Osstell device (Integration diagnostic Ltd. Company, Sävedalen, Sweden). Primary and secondary implant stability were analyzed and compared. The use of the Osstell and ISQ values were obtained by a blinded operator

SECONDARY OUTCOMES:
Radiographic assessment of the management of the crestal bone width and changes in labial bone thickness. | 4 months
  A postoperative CBCT will be taken within 24 hours of implant placement followed by a 6-months scan, and values will be compared with the preoperative record. The assessment will be conducted using the tools on the "On Demand 3D App." Software*. The following criteria will be assessed:

CONTACTS AND LOCATIONS:
Overall Officials: yehia El-Mahallawy, Phd, Principal Investigator — Faculty of Dentistry, Alexandria University, Alexandria, Alexandria
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP
Access Criteria: to any one who required them after deidentification